CLINICAL TRIAL: NCT01687127
Title: Metabolic Consequences of High-Dose Folic Acid Supplementation on Kinetics of 1-Carbon Metabolism
Brief Title: Impact of High-dose Folic Acid Supplementation on Pathways Linked to DNA Formation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Yvonne Lamers, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: H11-03009; CIHR Application Nr. 247226 (Other Grant/Funding Number: Canadian Institutes of Health Research - Application Nr. 247226)
Record Dates: First submitted 2012-09-13; First posted 2012-09-18 (Estimated); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: One-carbon Metabolism in Healthy Individuals
Keywords: folic acid; folate; 5-methyltetrahydrofolate; supplements; women; one-carbon metabolism; methionine; DNA methylation; in vivo kinetics
MeSH Terms: interventions — Folic Acid; Leucovorin; 5-methyltetrahydrofolate; levomefolate calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Folic acid supplementation (Experimental): Folic acid will be given orally in form of tablets. A supplement of 1 mg will be taken daily for 12 weeks. Thereafter, a supplement of 5 mg will be taken daily for 12 weeks (i.e., until Week 24). At baseline, Week 12, and Week 24, subjects will receive a 9-hour primed constant infusion of amino acids in saline solution for quantification of kinetics of one-carbon metabolism.
  Interventions: Dietary Supplement: Folic acid
- 5-MTHF supplementation (Experimental): The calcium salt of 5-methyltetrahydrofolate (5-MTHF; Brand name "Metafolin") will be given orally in form of tablets. A supplement of 1 mg will be taken daily for 12 weeks. Thereafter, a supplement of 5 mg will be taken daily for 12 weeks (i.e., until Week 24). At baseline, Week 12, and Week 24, subjects will receive a 9-hour primed constant infusion of amino acids in saline solution for quantification of kinetics of one-carbon metabolism.
  Interventions: Dietary Supplement: 5-methyltetrahydrofolate, calcium salt

INTERVENTIONS:
Dietary Supplement: Folic acid — Supplement
  Other Names: Pteroylmonoglutamic acid
  Arms: Folic acid supplementation
Dietary Supplement: 5-methyltetrahydrofolate, calcium salt — Supplement
  Other Names: 5-MTHF; Metafolin (brand name); Levomefolic acid
  Arms: 5-MTHF supplementation

SUMMARY:
Periconceptional supplementation with folic acid - the synthetic form of the B-vitamin folate - reduces the occurrence of adverse pregnancy outcomes such as spina bifida. The underlying biochemical mechanisms for how folic acid affects health outcomes however are unknown. The naturally occurring form 5-methyltetrahydrofolate (5-MTHF) is now available and discussed as an adequate substitute to folic acid. This study aims to determine the effect of folic acid compared to 5-MTHF on cellular mechanisms. Stable isotope tracer protocols will be used that allow determining the effect of folic acid on the dynamics of metabolic pathways in the human body.

Hypothesis: Supplementation with high-dose folic acid alters the turnover rate of folate dependent pathways in healthy humans; but 5-MTHF does not. Genetic variations in a key enzyme of the folate metabolism will aggravate the effect of folic acid on the metabolic pathways.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy
* Body mass index of between 19-24 kg/m2
* Normal folate, vitamin B12, and B6 status

Exclusion Criteria:

* Unable to swallow tablets
* Unable to receive intravenous catheters
* Use of vitamin supplements, amino acid or protein supplements for more than six months before study participation
* Chronic consumption of a high-protein diet (e.g. Atkins Diet)
* Medical conditions such as diabetes, asthma, cancer, cardiovascular disease, a history of neural tube defect (such as spina bifida) affected pregnancy, have had gastrointestinal surgery, abnormal kidney, thyroid function, or psychiatric illness, or any other chronic disease
* Pregnancy or lactation
* Smoking, use of recreational drugs, and/or consumption of more than one alcohol drink per day or more than seven per week.
* Use of long-term prescription medication such as hormonal contraceptives, antidepressants, anticonvulsants, anticoagulants, or other chronic medication
* Blood donation in the last three months prior to study start
* Unable to provide informed consent, or unable to read and write English
* Low compliance to intervention as determined by early steady-state or reduction in blood folate concentrations

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Plateau enrichment of infused amino acid tracers and related metabolites to quantify turnover rates of folate dependent pathways | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Lamers, PhD, Principal Investigator — University of British Columbia
Locations (1):
- Children's and Women's Health Centre of BC (incl. Sunny Hill), Child and Family Research Institute, Vancouver, British Columbia, Canada